CLINICAL TRIAL: NCT05792618
Title: Stroke Patients and Family in Rural China: A Longitudinal Study in Hebei Province
Brief Title: Stroke Patients and Family Longitudinal Study in Rural China
Acronym: SaFaRI
Status: Completed | Type: Observational
Sponsor: Duke Kunshan University (Other)
Collaborators: Peking Union Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: 2022DKU
Record Dates: First submitted 2022-11-14; First posted 2023-03-31 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SaFaRI is a large prospective cohort study in Hebei Province, rural Northern China including 1,299 stroke patients and their spouses. Follow-up visits take place from baseline until the fifth year after the baseline survey, investigating the lifestyle and health behavior, disease history, medication and adherence to medication, health status and self-reported health, cognitive function, and medication cost. As additional measures, the investigators will collect information on hospitalization, recurrence, and vital status from county medical insurance system and death record system. Patients will also have a physical examination comprising of assessment of blood pressure, weight, height, waist circumference, neck circumference, grip strength and the "Timed Up and Go" test.

DETAILED DESCRIPTION:
SaFaRI is a prospective longitudinal follow-up study based on a cluster-randomized controlled trial (System-integrated technology-enabled model of care to improve the health of stroke patients in rural China, SINEMA study) to evaluate the effectiveness of the SINEMA model to improve the secondary prevention of stroke in Nanhe County, a rural area of Hebei Province, China. A total of 1299 stroke patients were included at baseline, of which 25 villages received the SINEMA intervention package.

TThe SaFaRI study conducted a new follow-up round for participants of the SINEMA trial in 2023. Initially including 1299 stroke patients at baseline, this follow-up also encompassed the patients' spouses. The study aimed to: 1) Evaluate the stroke patients' blood pressure reduction, adherence to secondary prevention medications, physical activity, recurrence of stroke, hospitalization rates, and mortality. 2) Assess the long-term effectiveness of the SINEMA intervention model after a 5-year follow-up by examining the knowledge, attitudes, and practices of village doctors. 3) Establish a dynamic and continuous cohort of stroke patients, representative of northern rural China, using data from the baseline and the 1-year follow-up visits.

In 2024, the cohort underwent another follow-up, which expanded to include the collection of additional diseases and their diagnosis dates, and also surveyed patients regarding their sensory and viatality function.

ELIGIBILITY:
The eligible stroke patients should meet all the following criteria: those who

* aged more than 18 years old
* have a history of stroke diagnosed at county or higher-level hospitals, and are in stable condition;
* have at least a basic communication ability;
* give their informed consent and are willing to participate in the study.
* have participated in the primary care-based integrated mobile health intervention for stroke management in rural China (SINEMA).

And excluding those who

* have serious mental diseases;
* have other serious diseases, and have a remaining life expectancy of less than 6 months.

The eligible spouses should meet all the following criteria: those who

* aged more than 18 years old
* is the spouse of the stroke patient who participates in SINEMA study;
* have at least a basic communication ability;
* give their informed consent and are willing to participate in the study.

And excluding those who

* have serious mental diseases;
* have other serious diseases, and have a remaining life expectancy of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from the SENEMA study sample and their spouses. The SENEMA study sample has the following characteristics: over 18 years old, have a history of stroke diagnosed at county hospital or higher-level facilities, are currently in a clinically stable condition and not receiving acute stroke treatment, will live in this village for at least 9 months during the next 12 months, have basic communication ability and give their informed consent. A total of 1299 individuals were included at baseline. After excluding those who died during the 1-year follow-up (n = 30), a total of 1269 people will be included in the 5-year follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 1299 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | change from baseline to follow-up
  change in blood pressure
Weight | change from baseline to follow-up
  change in weight
Height | change from baseline to follow-up
  change in height
Grip strength | at various follow-up stages
  Grip strength (kilogram) will be estimated through the dynamometer (YuejianTM WL-1000, Nantong, China). Trained examiners will instruct people to hold the dynamometer and squeeze the handle for a few seconds. This study both measures right and left-hand grip strength twice in each hand. The grip strength will be recorded separately. If the average grip strength of both right and left hand of is all less than the criteria (man < 30 kg, woman < 20 kg), it is defined as weak grip strength.
Neck circumference | at various follow-up stages
  participants' neck circumference
Waist circumference | at various follow-up stages
  Participants' waist circumference
Mobility | at various follow-up stages
  measured by timed-up-and-go test, a simple and quick functional mobility test that requires the participants to stand up, walk 3 meters, turn, walk back, and sit down

SECONDARY OUTCOMES:
Cognitive function | at various follow-up stages
  measured by a brief version of the Community Screening Instrument for Dementia (CSI-D). The brief CSI-D was developed by Martin Prince, which consist of 7 cognitive items (Prince, M., Acosta, D., Ferri, C. P., Guerra, M., Huang, Y., Jacob, K. S., ... & 10/66 Dementia Group. (2011). A brief dementia screener suitable for use by non-specialists in resource poor settings-the cross-cultural derivation and validation of the brief Community Screening Instrument for Dementia. International journal of geriatric psychiatry, 26(9), 899-907.). The score of the brief CSI-D ranges from 0 to 9, with 0-4 represent Probable dementia, 5-6 represent Possible dementia, and 7-9 represent Normal.
Mental Health | change from baseline to follow-up
  measured by using Patient Health Questions-9, an international standard instrument for screening, monitoring and measuring the severity of depression. The total scores range from 0 (no depression) to 27 (severe depression).
Health related quality of life | change from baseline to follow-up
  measured using EuroQol-5 Dimensions-5L (EQ5D-5L). EQ-5D-5L descriptive system comprises the following five dimensions, each describing a different aspect of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. For each domain, the total scores range from 0 (indicating no problem) to 5 (indicating unable to/extreme problems). In addition, the participants were required to assess how their health is today by write a number from 0 to 100 on the numbered scale. 100 means the best health the participant can image, 0 means the worst health the participant can image.
Medication adherence | change from baseline to follow-up
  measured using 4 item Morisky Green Levine Scale-4 (MMAS-4), which scores adherence from 0-4 and continuation of medication taking is measured by the total months of medication taking
Disease history | change from baseline to follow-up
  collected through questionnaire and medical insurance records
Lifestyle risk factors | change from baseline to follow-up
  The factors include lack of exercise, alcohol, diet, obesity, and smoking, and will be collected through questionnaire.
Basic activities of daily living | at various follow-up stages
  measured by the basic activities of daily living (ADL). The basic ADL include the following categories: Ambulating, Feeding, Dressing, Personal hygiene, Continence, and Toileting. The ADL score ranges from 0 to 12. Limitation in ADL was defined as being scored greater than 0 on ADL scales, i.e., having some or severe limitation in at least one ADL item. Higher scores mean a worse functional independence.
Instrumental activities of daily living | at various follow-up stages
  measured by the Lawton Instrumental Activities of Daily Living (IADL) Scale to evaluate independent living skills. The scale measures eight domains of function, including food preparation, housekeeping, laundering. The IADL score ranges from 0 to 14. Limitation in IADL was defined as being scored greater than 0 on IADL scales, i.e., having some or severe limitation in at least one IADL item. Higher scores mean a worse functional independence.
Disability | change from baseline to follow-up
  measured using modified Rankin Scale (ranged 0 (no symptom) to 5 severe disability)
Multimorbidity | at various follow-up stages
  Assessed by determining whether participants had additional diseases diagnosed in the hospital, excluding stroke
Sensory and vitality functions | at various follow-up stages
  Assessed by querying your usual use of corrective lenses for vision, your ability to recognize distant and close objects, your use of hearing aids, and the quality of your hearing in different conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanhe County, Xingtai, Hebei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang B, Gong E, Chen X, Tan J, Peoples N, Li Y, Cai J, Li Y, Oldenburg B, Chen C, Dong D, Zhang X, Finkelstein E, Si L, Yan LL. Economic Evaluation of a Multicomponent mHealth Intervention for Stroke Management in Rural China: Cluster-Randomized Trial With 6-Year Follow-Up. JMIR Mhealth Uhealth. 2025 Sep 11;13:e75326. doi: 10.2196/75326. PMID 40934495
- [Derived] Tan J, Gong E, Gallis JA, Sun S, Chen X, Turner EL, Luo S, Duan J, Li Z, Wang Y, Yang B, Lu S, Tang S, Bettger JP, Oldenburg B, Miranda JJ, Karmacharya B, Kinra S, Shao R, Ebrahim S, Yan LL. Primary Care-Based Digital Health-Enabled Stroke Management Intervention: Long-Term Follow-Up of a Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2449561. doi: 10.1001/jamanetworkopen.2024.49561. PMID 39671199